CLINICAL TRIAL: NCT03803800
Title: Periodized Rehabilitation and Beta-alanine Supplementation in Multiple Sclerosis
Acronym: MSCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Prof. Dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16.111/REVA16.14
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Periodized exercise therapy; Ergogenic supplementation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Congresses as Topic; beta-Alanine

STUDY DESIGN:
Intervention Model Description: Four intervention groups following either 12 weeks of 'classical' moderate intensity cardiovascular exercise therapy (n=40) or periodized exercise therapy (n=40), with (MSβclassic, n=20; MSβperiod, n=20) or without (MSclassic, n=20; MSperiod, n=20) β-alanine supplementation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects involved (participants, care providor, asessor) are blinded to the supplementation (beta-alanine vs placebo).
  Outcome assessors are blinded to the exercise intervention (classic vs periodized training)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Classic training & beta-alanine (Experimental): Subjects following 12 weeks of classic, progressive endurance training, with the addition of ergogenic supplements (beta-alanine supplementation).
  Interventions: Other: Classic, progressive endurance training; Dietary Supplement: beta-alanine
- Classic training & placebo (Placebo Comparator): Subjects following 12 weeks of classic, progressive endurance training, without the addition of ergogenic supplements (placebo supplements).
  Interventions: Other: Classic, progressive endurance training
- Periodized training & beta-alanine (Experimental): Subjects following 12 weeks of periodized exercise training, with the addition of ergogenic supplements (beta-alanine supplementation).
  Interventions: Other: Periodized exercise training; Dietary Supplement: beta-alanine
- Periodized training & placebo (Placebo Comparator): Subjects following 12 weeks of periodized exercise training, without the addition of ergogenic supplements (placebo supplements).
  Interventions: Other: Periodized exercise training

INTERVENTIONS:
Other: Classic, progressive endurance training — Moderate intensity endurance training will be performed following a sequence of 5 training sessions every 2 weeks throughout the 12-week intervention. Sessions will include 60min of cycling on a stationary bicycle. Exercise intensity will match 60-80% of the maximal heart rate (HRmax)
  Arms: Classic training & beta-alanine; Classic training & placebo
Other: Periodized exercise training — Throughout the 12-week periodized intervention, subjects will perform four recurrent 3-week cycles of moderate endurance training (week 1,three sessions, 60min/session, 60-80% HRmax), high intensity interval training (week 2, three sessions, 10min/session, 3x20sec supramaximal sprint interspersed with recovery intervals of 2min), and recovery weeks (week 3, one high intense interval session as described above)
  Arms: Periodized training & beta-alanine; Periodized training & placebo
Dietary Supplement: beta-alanine — Some subjects will receive the ergogenic supplement beta-alanine.
  Arms: Classic training & beta-alanine; Periodized training & beta-alanine

SUMMARY:
Exercise therapy and increased physical activity in persons with Multiple Sclerosis (MS) improves mobility, muscular strength, physical fitness and fatigue without increasing relapse rate. As such, physical activity and more particular exercise therapy have become an important part of MS rehabilitation. Despite the fact that the positive effects of exercise therapy in MS are obvious only 43 percent of the MS community reports to participate in an exercise program4. Therefore, new exercise therapy approaches that further optimize rehabilitation, improve exercise adherence and promote participation in physical exercise in MS are interesting to explore. Therefore, the randomized controlled trial investigates two types of exercise interventions (classic progressive vs periodized) with or without the addition of ergogenic supplements (beta-alanine vs placebo).

DETAILED DESCRIPTION:
Following inclusion, baseline measurements (PRE) will be performed in MS patients (n=80). First, static(isometric) muscle strength (dynamometry), exercise capacity (maximal graded exercise test) and body composition (DEXA) will be evaluated. After 4 days of recovery, m. vastus lateralis muscle samples (Bergström procedure) will be taken. Hereafter, MS patients will be randomly allocated to one of four intervention groups following either 12 weeks of 'classical' moderate intensity cardiovascular exercise therapy (n=40) or periodized exercise therapy (n=40), with (MSβclassic, n=20; MSβperiod, n=20) or without (MSclassic, n=20; MSperiod, n=20) β-alanine supplementation. Groups not receiving β-alanine supplements, will receive placebo tablets that will be identical in taste and appearance. To evaluate post training fatigue, perceived exertion will be recorded following each training session (6-20 BORG scale). Following 12 weeks of classic or periodized training POST intervention measurements will be performed similar to baseline.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis Multiple Sclerosis.
* Healthy control.
* Aged >18y.
* Written informed consent.

Exclusion criteria:

* Contraindications to perform moderate to high intensity exercise.
* Participation in another study.
* Experienced acute MS related exacerbation <6 months prior to start of the study
* EDSS score > 6

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 3 weeks
  Exercise capacity will be assessed using a maximal (12-lead ECG) graded cardiopulmonary exercise test (♂: 30W+15W/min, ♀: 20W+10W/min, GE eBike Basic®) with pulmonary gas exchange analysis (Jaeger Oxycon®). VO2, VE, RER will be monitored. This test will be performed at least 48 hours separated from the muscle strength test, to prevent interference of muscle fatigue. RER values will be evaluated to verify if the test was performed maximally (RER >1.1).
Serum lactate | 3 weeks
  During the exercise test, 2min capillary blood samples will be obtained to analyse blood lactate concentrations (Analox®) and determine the anaerobic threshold before, during and after exercise.
Body composition | 3 weeks
  hole body fat and lean tissue mass will be obtained using Dual Energy X-ray Absorptiometry scan (DEXA) (Hologic Series Delphi-A Fan Beam X-ray Bone Densitometer, Vilvoorde, Belgium).
Body mass index | 3 weeks
  Weight (calibrated analogue weight scale) and height will be combined to report BMI in kg/m^2.
Strength measurement | 3 weeks
  Quadriceps and hamstrings muscle strength will be assessed using a isokinetic dynamometer. Back- and abdominal muscle strength will be assessed using an isokinetic dynamometer (System 3, Biodex, ENRAF-NONIUS, New York, USA). After adequate warming-up and movement familiarization, subjects will perform 3 maximal isometric contractions of back- and abdominal muscles for 4-5sec. This test will be executed in two starting positions (semi-flexed and lumbar isolated) to evaluate adequate co-contraction of m.Iliopsoas and m.Glutei during back flexion and extension respectively.
Muscle carnosine concentration | 3 weeks
  Muscle biopsies will be obtained from the middle part of the m.vastus lateralis (Bergström needle technique), by an experienced medical doctor.. The first two samples will be immediately embedded in Tissue-Tek, frozen in isopentane cooled with liquid nitrogen and stored at -80°C, until further analysis will be performed. The second two samples will be 'snap freezed' between pincers cooled with liquid nitrogen, and also stored at -80°C until further analysis.
  Carnosine concentrations will be determined using high-performance liquid chromatography (HPLC). Samples (15mg) are deproteinized using 35% sulfosalicylic acid and centrifuged (5min, 16,000g). Deproteinized supernatant is mixed with AccQ Fluor Borate buffer and reconstituted Fluor Reagent (1:7:2) from the AccQTag chemistry kit (Waters). Derivatized samples are applied to a Waters HPLC system comprised of an AccQTag column (3.9x150mm) and fluorescence detector (excitation/emission wavelength: 250/395nm).

CONTACTS AND LOCATIONS:
Overall Officials: Bert O Eijnde, Principal Investigator — University Hasselt
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium